CLINICAL TRIAL: NCT05915104
Title: Efficacy and Safety of Budesonide MMX® vs. Budesonide CR for Induction of Remission in Microscopic Colitis: A Prospective, Randomized, Active Comparator Pilot Study
Brief Title: Efficacy and Safety of Budesonide MMX® vs. Budesonide CR for Induction of Remission in Microscopic Colitis
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of Calgary (Other)
Collaborators: Ferring Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: REB22-1240
Record Dates: First submitted 2023-06-13; First posted 2023-06-22 (Actual); Last update posted 2023-12-04 (Actual); Status verified 2023-06

CONDITIONS: Microscopic Colitis
MeSH Terms: conditions — Colitis, Microscopic | interventions — Capsules; Budesonide

STUDY DESIGN:
Intervention Model Description: This phase 2a trial is a prospective, randomized, single-blinded (investigator-blinded), active comparator clinical study. Eligible participants with active Microscopic Colitis will be randomized 1:1 to receive either budesonide MMX® or budesonide CR 9 mg daily for 8 weeks.
Who Masked: Investigator, Outcomes Assessor
Masking Description: All qualified participants will be randomly assigned in a 1:1 ratio to receive budesonide MMX® or budesonide CR. Blocked randomization (block size of 8) will be stratified on disease subtype (collagenous colitis vs. lymphocytic colitis). Randomization will be conducted through the REDCap® clinical trials randomization module, which will generate a random, blinded allocation sequence that will be concealed to both investigators and participants.
  An independent pharmacist will prepare all treatment packages. Budesonide will be packaged into 4-week increments (two packages per 8-week treatment course). These treatment packages will be identical in appearance and size and labelled with a randomly generated study identification number. Investigators will not know the contents of each treatment package.
  At the randomization visit, eligible participants will be randomized and be given the corresponding treatment package. Participants will not be blinded to treatment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Budesonide MMX® (Experimental): Participant received 9 mg delayed and extended-release tablet, once daily, oral administration, for 8 weeks
  Interventions: Drug: Budesonide MMX®
- Budesonide controlled ileal release (CR) capsules (Active Comparator): Participant received three 3 mg capsules, daily oral administration, for 8 weeks
  Interventions: Drug: Budesonide controlled ileal release (CR) capsules

INTERVENTIONS:
Drug: Budesonide MMX® — 9 mg delayed and extended-release tablet once daily
  Other Names: Cortiment®
  Arms: Budesonide MMX®
Drug: Budesonide controlled ileal release (CR) capsules — three 3 mg capsules daily oral administration for 8 weeks
  Other Names: Entocort®
  Arms: Budesonide controlled ileal release (CR) capsules

SUMMARY:
The purpose of this research study is to compare how well two formulations of budesonide (budesonide MMX [Cortiment] and budesonide CR [Entocort]) work for treating patients with microscopic colitis.

DETAILED DESCRIPTION:
After being informed of the study and potential risks, patients with symptomatically active microscopic colitis who provide written informed consent will undergo a 4-week screening period to determine their eligibility for the study. At week 0, eligible patients will be randomized in a single blind manner (patients will be aware, while investigators will be blinded) in a 1:1 ratio to budesonide MMX (9mg once daily) or budesonide CR (3mg three times daily). The total treatment duration will be for 8 weeks. The primary outcome will be clinical remission, defined by the Hjortswang criteria (daily average <3 loose/watery bowel movements per 24 hours in the week preceding the final assessment (loose/watery stool consistency will be measured using the Bristol Stool Chart (types 6 and 7)).

ELIGIBILITY:
Inclusion Criteria:

* Male or non-pregnant, non-lactating females, 18-80 years old years of age
* Females of childbearing potential must be taking adequate contraceptive precautions (i.e., implants, injectables, hormonal intrauterine devices, combined hormonal contraceptives, having a vasectomized partner or total abstinence from heterosexual relations with no plans of becoming pregnant through insemination or in vitro fertilization) and have a negative urine pregnancy test prior to randomization.
* Active symptoms of MC defined by non-bloody, watery diarrhea or loose bowel movements for at least 12 weeks (for patients with newly diagnosed MC) or a history of clinical relapse for at least one week before randomization in patients with previously established MC, and with >=28 stools within 7 days preceding randomization, of which >=20 were watery/soft stools
* Colonoscopy or flexible sigmoidoscopy with histologically confirmed MC, defined by signs of inflammation of the lamina propria and either:
* lymphocytic colitis: ≥20 IELs/100 surface epithelial cells
* collagenous colitis: subepithelial collagen band >10 micrometers in diameter
* Ability of subject to participate fully in all aspects of this clinical trial
* Written informed consent must be obtained and documented

Exclusion Criteria:

* Evidence of infectious diarrhea (proved by stool culture or colonic biopsy), diarrhea due to other organic diseases of the gastrointestinal tract including Crohn's disease, ulcerative colitis, ischemic colitis, Celiac disease (ruled out by either duodenal biopsy or serum antibodies), radiation colitis, or polyps >2cm, suspicion of drug-induced MC
* History of partial or total colonic resection
* Previous exposure to >7 days of any budesonide formulation for treatment of MC
* Unwillingness to withhold protocol-proscribed medications during the trial
* Received any of: aminosalicylates, corticosteroids (other than budesonide), immunosuppressants (including thiopurines and methotrexate), bismuth subsalicylate, cholestyramine, biological treatments, or antibiotics (except for up to a 7-day course for conditions unrelated to microscopic colitis) within 8 weeks of randomization
* Use of loperamide or diphenoxylate/atropine as an anti-diarrheal agent is not permitted during the screening period
* Serious underlying disease other than MC which in the opinion of the investigator may interfere with the subject's ability to participate fully in the study, including a history of:
* Severe anaemia (haemoglobin < 90 g/L) or leukopenia (white blood cell count < 2.5 x 109 cells/L)
* Known infection with hepatitis B, hepatitis C, or human immunodeficiency virus not on effective anti-viral therapy
* Active malignancy
* Cirrhosis or significant hepatic or renal insufficiency
* Poorly controlled type 1 or type 2 diabetes
* Glaucoma
* History of alcohol or drug abuse which in the opinion of the investigator may interfere with the subject's ability to comply with the study procedures.
* Pregnant or lactating women
* Hypersensitivity to the active ingredient of budesonide MMX® or budesonide CR and excipients

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2024-01-01 (Estimated); Primary Completion 2026-09-01 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Clinical remission | Week 8
  Hjortswang criteria defines clinical remission as a daily average <3 loose/watery bowel movements per 24 hours in the week preceding the final assessment (loose/watery stool consistency will be measured using the Bristol Stool Chart (types 6 and 7)

SECONDARY OUTCOMES:
Histologic remission | Week 8
  <20 IELs/100 surface epithelial cells and subepithelial collagen band <10 micrometers in biopsy samples and a reduction in lamina propria inflammation
Histologic response | Week 8
  50% reduction in IEL count or subepithelial collagen band thickness compared to baseline and/or a reduction in lamina propria inflammation
Clinical response | Week 8
  50% reduction in average daily stool frequency for the week prior to final assessment compared to baseline
Patient-reported symptom improvement | Week 8
  Change in the European Microscopic Colitis Activity Index (E-MCAI) and its component items, including stool frequency and consistency (stools per day, solid vs. loose stools, stools of each Bristol Stool chart consistency), stools at night, feeling of a need to pass more stools shortly after a bowel movement, urgency of defecation, leakage, and abdominal pain

CONTACTS AND LOCATIONS:
Overall Officials: Christopher Ma, MD MPH, Principal Investigator — University of Calgary

IPD SHARING:
Plan to Share IPD: Yes
Deidentified IPD may be shared upon completion of the study and with formal written request
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Data will be available and stored for 15 years after the study completion